CLINICAL TRIAL: NCT06269991
Title: Investigation of the Effects of Facial Anthropometric Measurements and Anthropometry Related Parameters on Sports Performance in Archers
Brief Title: Fascial Anthropometry in Archery Athletes
Status: Not yet recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aynur Demirel, PT, PhD, Assoc. Prof., Hacettepe University
Other Study IDs: SBA23/083
Record Dates: First submitted 2023-12-28; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Sports Physical Therapy
Keywords: athletes; anthropometry; somatotypes; archery; posture; athletic performance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- bow category: the athletes using recurve bow or compound bow will investigating.

SUMMARY:
In archery, the body morphological and anthropometric characteristics of the prominent athletes change. It is important to examine facial anthropometry, especially since the athlete's equipment touches the facial area, and there are no studies on this subject. The aim of this study is to determine the relationship between facial anthropometric measurements and anthropometry-related parameters and sports performance in archery athletes.

DETAILED DESCRIPTION:
Within the scope of the study, a total of at least 60 athletes, between the ages of 9-18, who have been training archery at least twice a week for at least 2 years, who have not changed their bow category since it started, who do not have a temporomandibular joint problem, and who volunteer to participate in the study, will be recruited in equal numbers from each age category. Within the scope of evaluation; Demographic information and features regarding archery equipment will be recorded. Within the scope of anthropometric measurements; adipose tissue measurements with skinfold; circumference measurements and length measurements with tape measure; diameter measurements with caliper; Facial anthropometric measurements will be measured with a caliper/tape measure. Formulary named "Heath-Carter Anthropometric Somatotype Technique" to determine the body somatotypes of athletes; Lateral photography for biomechanical evaluation of the craniocervical region; Hand Grip Strength Test for performance evaluation; Corbin Postural Assessment Scale will be used for posture evaluation. In order to determine the shooting performance, the athletes' actual competition scores in the last year will be recorded. Medicine ball throwing test, upper extremity y balance test and closed kinetic chain upper extremity stability test will be used to evaluate upper extremity performance. For statistical analysis, normal distribution of parameters will be examined. To determine the relationship between shooting performance and stabilization and related parameters, Pearson test will be used for normally distributed parameters and Spearman correlation test will be used for non-normally distributed parameters.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 9-18 years.
* Having been practicing archery at least twice a week for at least 2 years.
* Not having changed the bow category since it started.
* Fonseca Anamnestic Questionnaire result is between 0-15 points
* volunteering to participate in the study

Exclusion Criteria:

* Having had surgery involving the spine and upper extremities in the last year
* Scoliosis being diagnosed
* Having an orthopedic, neurological or musculoskeletal disease that involves the upper extremity and prevents shooting
* Having received orthodontic treatment
* orthodontic surgery to have had
* Being actively involved in another sports branch for at least 1 year

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: being archer at least two years.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2024-09-06 (Estimated); Study Completion 2025-09-06 (Estimated)

PRIMARY OUTCOMES:
evaluation of cervical region biomechanic | baseline
  Angle evaluation via photographic analysis
fat tissue distribution | baseline
  Fat tissue distribution will measure via skinfold in Triceps, subscapular, suprailiac regions.
head circumference | baseline
  Head circumference will measure around the head via tape.
extremity circumference | baseline
  arm and leg circumference will measure with a tape measure around the mid-way point between the proximal and distal joints of the athletes and will record in centimeter.
extremity lengt measurement | baseline
  upper and lower extremity lenght will measure via tape and will record in centimeter.
knee and elbow diameter | baseline
  knee and elbow diameter will measure via caliper.
nose width | baseline
  the width will measure via caliper.
chin width | baseline
  the width will measure via caliper.
face width | baseline
  the width will measure via caliper.
head width | baseline
  the width will measure via caliper.
nose protrusion | baseline
  the protrusion will measure via caliper.
nose lenght | baseline
  the lenght will measure via caliper.
head lenght | baseline
  the lenght will measure via caliper.
face lenght | baseline
  the lenght will measure via caliper.
lip lenght | baseline
  the lenght will measure via caliper.

SECONDARY OUTCOMES:
Assessment of Perıpheral Muscle Strength | baseline
  peripheral muscle strength will assessvia jamar hand dynamometer
postural analysis | baseline
  Posture will analyse via corbin postural assessment scale
Evaluation of shooting performance | baseline
  competition scores will record as shooting performance
The seated medicine ball throw (SMBT) | baseline
  This test is a field test intended to assess upper-body muscular power by measuring the maximal distance an individual can throw a medicine ball from an isolated in seated position.
Closed Kinetic Chain Upper Extremity Stability Test | baseline
  The test consists in counting how much times, during 15 seconds, the subject assuming a push-up position is able to touch his/her supporting hand with the swinging hand
Upper Quarter Y Balance Test | baseline
  The test consisted of the subject reaching in the 3 reach directions (Medial, Superolateral, Inferolateral) with the free hand while maintaining a push-up position with feet shoulder width apart.

CONTACTS AND LOCATIONS:
Overall Officials: Aynur Demirel, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided